CLINICAL TRIAL: NCT00833378
Title: A Phase I, Open-label, Single Sequence, Crossover Study Evaluating the Safety and the Pharmacokinetics of Lopinavir/Ritonavir and Eltrombopag Given Alone and When Co-administered in Healthy Adult Subjects.
Brief Title: Drug Interaction Study Between Eltrombopag and Lopinavir/Ritonavir in Healthy Adult Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111716
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Hepatitis C
Keywords: Drug interaction, SB-497115 (eltrombopag), Kaletra (Lopinavir, Ritonavir),thrombocytopenia, pharmacokinetics
MeSH Terms: conditions — Hepatitis C | interventions — eltrombopag; Lopinavir; Ritonavir

ARMS (3):
- Period 2 (Active Comparator): Treatment B
  Interventions: Drug: Lopinavir/Ritonavir
- Period 1 (Active Comparator): Treatment A
  Interventions: Drug: Eltrombopag
- Period 3 (Active Comparator): Treatment C
  Interventions: Drug: Eltrombopag and Lopinavir/Ritonavir

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag 100 mg single oral dose
  Arms: Period 1
Drug: Lopinavir/Ritonavir — Lopinavir/Ritonavir 400/100 mg oral dose given twice a day for 14 days
  Arms: Period 2
Drug: Eltrombopag and Lopinavir/Ritonavir — Elrombopag 100 mg single oral dose and Lopinavir/Ritonavir 400/100 mg oral dose given in the AM and PM
  Arms: Period 3

SUMMARY:
This is a Phase I, open-label, single sequence, crossover study to be conducted in healthy adult subjects. There will be a screening visit, three treatment periods, and a follow-up visit. In Period 1, subjects will receive a single dose of eltrombopag on Day 1, and PK sampling will occur for 72 hours. In Period 2, subjects will receive LPV/RTV for 14 days with PK sampling for 12 hours. In Period 3, subjects will receive a single dose of eltrombopag with LPV/RTV on Day 1 only with PK sampling for 72 hours. Subjects will return for a follow-up visit within 10 to 14 days of the last dose of study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no clinically significant abnormality identified by physician by evaluation of medical history, physical examination, clinical laboratory tests or electrocardiogram (ECG).
* Able to swallow and retain oral medication.
* Male and female subjects between the ages of 18 to 64 years of age inclusive, at the time of signing the informed consent.
* Subject is able to understand and comply with the protocol requirements, instructions and restrictions.
* Capable of giving written informed consent which includes compliance with the requirements and restrictions listed in the consent form. Signed informed consent must be on file prior to screening procedures.
* Body weight ≥ 50kg (110 lbs) for men and ≥ 45 kg (99 lbs) for women and body mass index (BMI) of 18.5 to 29.9 kg/m2 inclusive.
* Male subjects, who are not surgically sterile, must agree on abstinence or to use a double barrier method, such as, a condom plus spermicidal agent (foam/gel/film/cream/suppository). This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of medication.-
* A female subject is eligible to participate if she is neither pregnant nor lactating, and falls into one of the following categories:

  * non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or bilateral oophorectomy, or postmenopausal females defined as being amenorrheic for greater than 1 year and having serum estradiol and follicle stimulating hormone levels consistent with menopause.
  * child-bearing potential with negative β human chorionic gonadotropin (βhCG) test and agrees to comply with recognized non-hormonal contraceptive methods from screening or at least two weeks prior to first dose (whichever is earlier) until the follow-up visit. Recognized non-hormonal contraceptive methods include: complete abstinence from intercourse, two forms of barrier contraception (e.g. condom with spermicide, or diaphragm with spermicide), or intrauterine device (IUD).

Exclusion Criteria:

* History of Gilbert's syndrome.
* Any previous history of deep vein thrombosis or any other thromboembolic event. 3. History of thrombocytopenia or bleeding due to abnormal platelet number or function. 4. Clotting factor abnormalities associated with hypercoagulability, specifically Factor V Leiden, Protein C or Protein S deficiency or antithrombin III deficiency. 5. Elevated blood pressure (BP) at screening (systolic >140 mm Hg, diastolic >85 mm Hg). If the subject's BP is elevated on the first measurement, complete two additional BP measurements 2 minutes apart and average the three assessments to evaluate this criteria. If averaged BP exceeds the safety criteria, the subject should be excluded.

  6. History of atrial fibrillation, mitral valve prolapse, significant heart murmur or vascular bruit. 7. Prolonged QTc interval (Bazett's) at screening (for females > 450 msec and for males > 430 msec). If the QTc interval is prolonged on the initial ECG, then complete two additional ECGs 5 minutes apart and take the average QTc measurements of all three ECGs to evaluate this criteria. If averaged QTc exceeds the safety criteria, the subject should be excluded. 8. Female subjects currently receiving hormone replacement therapy (HRT). 9. Positive for HIV, hepatitis B virus or hepatitis C virus assays at screening.

  10. Positive urine drug screen including alcohol at screening or pre-dose (Day -1).

  11. History of alcohol/drug abuse or dependence within 12 months of the study. RM2008/00650/00 CONFIDENTIAL TPL111716 25 CONFIDENTIAL RM2008/00650/00 TPL111716 26 12. History of alcohol consumption in the past six months exceeding 7 units/week for women and 14 units/week for men (where 1 unit = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor). 13. Urinary cotinine levels indicative of smoking at screening or pre-dose (Day -1).

History of regular use of tobacco- or nicotine-containing products within 6 months prior to screening. 14. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication. 15. Exposure to more than four new chemical entities within 12 months prior to the first dosing day. 16. Use of prescription or non-prescription drugs (including aspirin and non-steroidal anti-inflammatory drugs [NSAIDs]), vitamins, herbal and dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer, such as St. John's Wort) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety. 17. Subjects who have donated plasma within 7 days prior to the screening visit or where participation in this study would result in donation of blood in excess of 500 mL within a 56-day period. 18. History of sensitivity to any of the study medications, or components thereof.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01-19 (Actual); Primary Completion 2009-03-11 (Actual); Study Completion 2009-03-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters per the protocol | sixteen days

SECONDARY OUTCOMES:
Safety parameters including vital signs, laboratory assessments, ECG measurements and adverse events reporting | sixteen days of treatment and follow-up period.
Pharmacokinetic parameters per the protocol | sixteen days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Buffalo, New York, United States

REFERENCES:
- [Background] Wire MB, McLean HB, Pendry C, Theodore D, Park JW, Peng B. Assessment of the pharmacokinetic interaction between eltrombopag and lopinavir-ritonavir in healthy adult subjects. Antimicrob Agents Chemother. 2012 Jun;56(6):2846-51. doi: 10.1128/AAC.05214-11. Epub 2012 Mar 5. PMID 22391553
- See also: Results for study 111716 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111716?search=study&search_terms=111716#rs